CLINICAL TRIAL: NCT01388530
Title: An Eight-Week, Open Trial Pilot Investigation of Trigeminal Nerve Stimulation for Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Trigeminal Nerve Stimulation for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: NeuroSigma, Inc. (Industry)
Responsible Party: Principal Investigator, James McGough, Professor of Clinical Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLA-TNS/ADHD
Record Dates: First submitted 2011-06-24; First posted 2011-07-06 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trigeminal nerve stimulation (Experimental): Open label treatment with trigeminal nerve stimulation in an 8-week trial.
  Interventions: Device: EMS 7500 Digital Muscle Stimulator

INTERVENTIONS:
Device: EMS 7500 Digital Muscle Stimulator — A standard FDA approved transcutaneous electrical nerve stimulation (TENS) unit will be used to apply low intensity stimulation to the trigeminal nerves during sleep.

SUMMARY:
This proposal seeks to obtain preliminary data on the potential efficacy, tolerability, and feasibility of trigeminal nerve stimulation (TNS) as a treatment for Attention-Deficit/Hyperactivity Disorder (ADHD). If successful, this open-label, exploratory, pilot study will provide a basis for a federal grant application and larger controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* male and female youth age 9 to 14 years with Diagnostic and Statistical Manuel -IV (DSM-IV) ADHD, combined subtype as determined by Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS) and clinical interview
* minimum scores of 12 on both the inattentive and hyperactive/impulsive subscales of the baseline ADHD-Rating Scale (ADHD-RS)S
* Clinical Global Impression- Severity (CGI-S) score at baseline
* no current medications with central nervous system (CNS) affects
* parents able and willing to monitor proper use of the stimulation device and complete all required rating scales.

Exclusion Criteria:

* impaired functioning to a degree that requires immediate initiation of ADHD medication in the opinion of the parents and/or investigator; 2) current diagnosis of pervasive developmental disorder or major depression.
* history of lifetime psychosis or mania
* current suicidality
* history of seizure disorder, tic disorder, or head injury with loss of consciousness.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J McGough, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated in July 2011 and ended in October 2012. Participants self-identified or were referred from community providers in response to public advertisements.
Pre-assignment Details: Following informed permission/assent participants were assessed for eligibility and if meeting inclusion/exclusion criteria initiated 8 weeks of open-label Trigeminal Nerve Stimulation (TNS) treatment.
Groups:
- Trigeminal Nerve Stimulation: Open label treatment with trigeminal nerve stimulation in an 8-week trial.
  EMS 7500 Digital Muscle Stimulator : A standard FDA approved transcutaneous electrical nerve stimulation (TENS) unit will be used to apply low intensity stimulation to the trigeminal nerves during sleep.
Period: Overall Study
Arm/Group | Trigeminal Nerve Stimulation
Started | 25
Completed | 20
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Trigeminal Nerve Stimulation
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.14 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: ADHD-IV Rating Scale (ADHD-RS)
Description: A standard, frequently used, clinician completed measure of Diagnostic and Statistical Manual -IV (DSM-IV) ADHD symptoms.
  Scale ranges from 0 (best) to 54 (worst).
  Unit of Measure - units on a scale.
  Outcome value reflects change from baseline at endpoint (Week 8) in ADHD-RS.
Time Frame: Baseline and Week 8.
Population: Participants with data at baseline and week 4. We included participants who participated in 4 weeks of treatment, but change comparison is baseline vs. week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trigeminal Nerve Stimulation
Number analyzed (Participants) | 22
units on a scale | 32.6 (1.58)

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: A global measure of clinical improvement compared with baseline.
  A standard clinical trials rating scale with value from 1 (very much improved) to 7 (very much worse).
  Unit of measure - percentage improved based on CGI-I scores of 1 and 2 versus all others.
Time Frame: Week 8
Population: Participants with data at baseline and week 4. As with the ADHD-RS, we included participants with at least 4 weeks of treatment, but outcome was assessed at Visit 8 compared with baseline.
Measure: Number; unit: percentage of improved
Arm/Group | Trigeminal Nerve Stimulation
Number analyzed (Participants) | 22
percentage of improved | 67

3. Secondary Outcome: Conners Global Index - Parent
Description: A standard, parent completed measure of ADHD symptoms.
  Scale range from 0 (best) to 27 (worst).
  Unit of Measure - units on a scale.
  Outcome value reflects change from baseline at endpoint (Week 8).
Time Frame: Baseline and Week 8.
Population: Participants with data at baseline and week 4. We required 4 weeks treatment to include in analysis, but analysis is based on comparison of baseline and week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trigeminal Nerve Stimulation
Number analyzed (Participants) | 22
units on a scale | 19.6 (1.3)

4. Secondary Outcome: Attention Network Task - Incongruent Reaction Time
Description: Laboratory measure of response inhibition. The measure assessed the reaction time in milliseconds (ms) using the Attention Network Task (ANT), which is a computerized test designed to evaluate the efficiency of an attention network.
  Outcome measure represents a change from Baseline at Week 8 for the ANT - Incongruent reaction time. Lower reaction time is consider a better outcome.
Time Frame: Baseline and Week 8.
Population: Participants with data at baseline and week 4. We included participants who completed 4 weeks of treatment, but comparison is based on Week 8 vs. baseline.
Measure: Mean (Standard Deviation); unit: milliseconds (ms).
Arm/Group | Trigeminal Nerve Stimulation
Number analyzed (Participants) | 22
milliseconds (ms). | 902.9 (31.2)

ADVERSE EVENTS:
Arm/Group | Trigeminal Nerve Stimulation
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Early terminations were due to ambivalence about participation of social difficulties with compliance. No one left the study for adverse events or safety reasons. There were no clinically meaningful adverse events related to treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No